CLINICAL TRIAL: NCT01014598
Title: Phase I Study of Targeted Lung Chemotherapy in the Treatment of Metastatic Tumors
Brief Title: Cisplatin in Treating Patients With Stage IIIB-IV Non-small Cell Lung Cancer or Lung Metastasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 70005; NCI-2009-01604 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 70005 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Malignant Neoplasm in the Lung; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Adult Soft Tissue Sarcoma; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Sarcoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (cisplatin) (Experimental): Patients receive cisplatin intra-arterially via isolated lung suffusion over 2 hours. Beginning approximately 2 weeks later (6-8 weeks if indicated for patients with sarcoma undergoing surgery after cisplatin), patients receive standard chemotherapy regimen.
  Interventions: Drug: Cisplatin; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cisplatin — Given intra-arterially via isolated lung suffusion
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of cisplatin in treating patients with stage IIIB-IV non-small cell lung cancer or tumors that have spread from where they started to the lung (metastasis). Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving cisplatin directly into the arteries around the tumor may kill more tumor cells and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose and dose-limiting toxicities of cisplatin when delivered selectively by isolated lung suffusion to patients with any biopsy or cytologically proven resectable or unresectable primary or secondary malignancy in the lung.

SECONDARY OBJECTIVES:

I. To assess lung tissue levels of cisplatin after isolated lung suffusion as a function of the dose delivered.

II. To evaluate systemic and pulmonary artery concentrations of cisplatin during isolated lung suffusion.

OUTLINE: This is a dose-escalation study.

Patients receive cisplatin intra-arterially via isolated lung suffusion over 2 hours. Beginning approximately 2 weeks later (6-8 weeks if indicated for patients with sarcoma undergoing surgery after cisplatin), patients receive standard chemotherapy regimen.

After completion of study treatment, patients are followed up for at least 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Any biopsy or cytologically proven resectable or unresectable primary or secondary (metastatic) malignancy in the lung; this is defined as

  * Tumors whose only remaining residual deposits are confined to the lungs OR
  * Oligometastatic tumors with > 80% of measurable tumor volume in the target lung In both of the above situations, no clinical evidence of central nervous system (CNS) metastases can exist; oligometastatic disease is difficult to define but would, as a guideline, have only 1-4 loci of disease established in 1-2 organ systems outside the affected lung; exceptions to these guidelines can occur, particularly in cases where sites of metastatic disease are equivocal or so minute that it would not exceed 20% of tumor volume
* Unresectable stage IV non-small cell lung cancer (NSCLC)
* Unresectable stage IIIB NSCLC
* Resectable metastatic sarcoma to lung (thoracoscopically resectable)
* Other malignancies that meet the criteria
* Eastern Cooperative Oncology Group performance status 0-1
* No oxygen needs (oxygen use per standard established criteria for oxygen requirements)
* Modified Borg dyspnea scale < 5
* Six minute walk >= 50% of the expected distance; this will not be used as exclusion criteria if due to a reason other than respiratory per judgment of physician e.g., pain
* Ambulatory and resting oxygen (O2) saturation > 88%
* PPO (predicted post operative)* forced expiratory volume in one second (FEV1) >= 50% predicted

  * PPO values should be calculated for each patient
* PPO * diffusing capacity of the lung for carbon monoxide (DLCO) >= 50% predicted

  * PPO values should be calculated for each patient
* PPO * vital capacity >= 50% predicted

  * PPO values should be calculated for each patient
* Granulocytes > 1,500 ul
* Platelets >= 100,000 ul
* Patients must sign a study-specific consent form prior to registration
* Tumor anatomy must allow the isolated lung suffusion in the judgment of the principal investigator (PI)

Exclusion Criteria:

* Uncontrolled intercurrent disease
* Prior chemotherapy for proven metastatic disease within 4 weeks
* Evidence of pulmonary toxicity from previous or ongoing chemotherapy
* Creatinine > 1.5 mg/dL
* Liver enzymes > 2 times upper normal
* Uncontrolled congestive heart failure (in judgment of the PI)
* Optional: ejection fraction < 40% for clinical evidence of insufficient cardiac reserve (multi gated acquisition scan [MUGA] or echocardiogram [ECHO] will be done only if indicated in the judgment of the PI)
* Myocardial infarction or angina within past 6 months
* Contraindications to anticoagulation
* Hydration intolerance (e.g., uncontrolled congestive heart failure [CHF])
* Human immunodeficiency virus positive (HIV+) on antiretroviral therapy
* Pregnant or lactating
* Diffuse pulmonary fibrosis involving over 25% of the total lung parenchyma
* Previous radiation for thorax
* Metastatic sarcoma to lung that is not able to have tumors resected thoracoscopically
* Prior lung removal in the affected lung (would have decreased lung volume)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-12-04 (Actual); Primary Completion 2013-10-23 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Acute toxicity assessed using CTCAE version 4.0 | Within 7 days from lung infusion
Frequency of patients experiencing dose limiting toxicities (DLT) as well as non-DLT | Within 30 days of the procedure
  DLT is defined according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. A grade 3 or above adverse event shall be considered a DLT in this study if attributed to the isolated lung suffusion cisplatin dose.
Reversibility of all toxicities from this approach. | Up to 90 days from the start of lung infusion therapy

SECONDARY OUTCOMES:
Lung, systemic, and pulmonary artery concentrations of cisplatin | Before pulmonary artery release, at 15 minutes, and 1 hour
  Analysis of variance models with appropriate transformations of the variables, or nonparametric tests such as the Kruskal-Wallis test will be used as appropriate.
Pulmonary function test with diffusion capacity | Up to 30 days post-treatment
  Will be summarized with respect to the percentage of cisplatin given directly to the lung. Analysis of variance models with appropriate transformations of the variables, or nonparametric tests such as the Kruskal-Wallis test will be used as appropriate.
Split lung function test | Up to 30 days post-treatment
  Will be summarized with respect to the percentage of cisplatin given directly to the lung. Analysis of variance models with appropriate transformations of the variables, or nonparametric tests such as the Kruskal-Wallis test will be used as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Chukwumere Nwogu, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States